CLINICAL TRIAL: NCT04605796
Title: A Single-arm, Open-label, Multi-center Phase II Clinical Study to Evaluate the Safety and Efficacy of Toripalimab Injection (JS001) Combined With Bevacizumab as the First-line Therapy for Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-034-II-HCC
Record Dates: First submitted 2020-09-22; First posted 2020-10-28 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Experimental group:
  Toripalimab combined with Bevacizumab
  Interventions: Combination Product: Toripalimab combined with Bevacizumab

INTERVENTIONS:
Combination Product: Toripalimab combined with Bevacizumab — Experimental group:
  Toripalimab, 240mg, IV infusion, every 3 weeks (q3w). combined with Lenvatinib 15 mg/kg (IV infusion, every 3 weeks (q3w).. Continuous infusion, in a cycle of 3 weeks (21 days), until occurrence of termination event specified in the protocol.

SUMMARY:
This is an open-label, single-arm, national multicenter phase II clinical study to preliminarily observe and evaluate the efficacy and safety of Toripalimab combined with Bevacizumab as the first-line therapy for advanced HCC The study will use safety/tolerability and ORR as the primary study objectives and indicators, and plans to enroll about 50-60 patients.

ELIGIBILITY:
"The patients meeting all the following inclusion criteria can be enrolled in this study:

1. Age of 18-70 years (inclusive), male or female.
2. HCC diagnosed by histopathological examination or Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2017 Edition).
3. Stage B (middle stage) or C (late stage) HCC determined in accordance with Barcelona Clinic Liver Cancer staging system (BCLC stage). In case of stage B, the patient must be unsuitable for surgery and/or local therapy, or have progressive disease after surgery and/or local therapy, or refuse surgery and/or local therapy (special instruction and signature required).
4. No previous use of any systemic therapy or HCC.
5. Having ≥ 1 measurable lesion in accordance with RECISTv1.1.
6. Grade A Child-Pugh hepatic function, with no history of hepatic encephalopathy.
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 0-1.
8. Expected survival ≥12 weeks.
9. Adequate hematologic and end-organ function..
10. In case of HBsAg (+) and/or HBcAb (+), HBV DNA is required to be < 500 IU/mL, and it is required to continue the effective anti-HBV therapy that has been adopted in the full course, or start to use Entecavir or tenofovir in the full course during the study. HBV/HCV co-infected patients will be excluded. Patients with a history of HCV infection but with negative HCV RNA PCR results can be considered uninfected with HCV.
11. Female patients of childbearing potential must receive serum pregnancy test within 7 days before enrollment, have negative result, and agree to use reliable and effective contraceptive methods during the trial and within 60 days after the last dose of study drug. The male patients whose partners are women of childbearing potential must agree to use reliable and effective contraceptive methods during the trial and within 60 days after the last dose of study drug.
12. Being voluntary to participate in the study, sufficiently informed consent and signature of written informed consent form, with good compliance.

Patients can not be enrolled in the study if any one of the following criteria is fulfilled:

1. Known cholangiocellular carcinoma (ICC) or mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma and hepatic fibrolamellar carcinoma.
2. Malignant tumor except HCC in the past 5 years: however, localized tumor cured in the study is excluded, including cervical carcinoma in situ, skin basal cell carcinoma and carcinoma in situ of prostate.
3. Hepatic surgery and/or local therapy or treatment with investigational product for HCC within 4 weeks prior to enrollment; palliative therapy for bone metastatic lesion within 2 weeks prior to enrollment. Toxicity reaction induced by previous therapy (except alopecia) not recovered to ≤ grade 1 (NCI-CTCAE v5.0). Chinese medicine preparation with anti-liver cancer effect within 2 weeks prior to enrollment.
4. Uncontrolled pericardial effusion, uncontrolled pleural effusion or clinically obvious moderate peritoneal effusion at screening,
5. History of gastrointestinal hemorrhage within 6 months prior to enrollment; the patients with portal hypertension need to receive gastroscopy to exclude the patients with "red sign", if they are considered by investigators to have high risk for hemorrhage . The patient needs to be excluded if there is a history of "red sign" in gastroscopy.
6. Having ≥ grade 3 (NCI-CTCAE v5.0) gastrointestinal or non-gastrointestinal fistula at present.
7. Patients with cancer thrombus in the main trunk of portal vein (Vp4), or cancer thrombus in inferior vena cava should be excluded. However, the patients with cancer thrombus in the main trunk of portal vein but unobstructed branch of contralateral portal vein are allowed to be enrolled.
8. Previous history of serious cardiovascular and cerebrovascular diseases:
9. Having major bleeding and coagulation disorders or other obvious evidence on hemorrhagic tendency:
10. Medium to large surgical treatment within 4 weeks prior to enrollment, however, not including diagnostic biopsy.
11. Central nervous system metastasis.
12. Serious, uncured wound, active ulcer or untreated bone fracture.
13. Vaccination of live vaccine within 30 days prior to enrollment.
14. Active autoimmune diseases requiring systemic treatment (i.e., immunomodulatory drug, corticosteroid or immunosuppressant) in the past 2 years; however, replacement therapy (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency) will not be considered as systemic therapy and is allowed to be used, and enrollment is allowed.
15. History of clear interstitial lung disease or non-infectious pneumonia, unless induced by local radiotherapy; history of active tuberculosis.
16. Any serious acute and chronic infection requiring systemic antibacterial, antifungal or antiviral therapy at screening, not including viral hepatitis.
17. Known history of human immunodeficiency virus (HIV) infection.
18. Previously receiving allogeneic stem cell or solid organ transplantation.

20. Known history of serious allergy to any monoclonal antibody, anti-angiogenesis targeted drug.

"

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 2 years
  Frequency table will be used to summarize occurrence of each treatment-emergent AE
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 2 years
  Number and incidence of abnormal laboratory examinations by treatment group.
ORR | Up to 2 years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).

SECONDARY OUTCOMES:
DoR | Up to 2 years
  The time from the first assessment of CR or PR to the first assessment of PD or death due to any cause.
DCR | Up to 2 years
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
TTP | Up to 2 years
  time from the start of treatment to progression of diease.
PFS | Up to 2 years
  PFS is defined as time from the start of treatment to progression of disease or death.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as time from the start of treatment until death due to any reason.

OTHER OUTCOMES:
PD-L1 | Up to 2 years
  Correlation between PD-L1 expression level in tumor tissue, proportion of strong positive expression of PD-L1
TMB | Up to 2 years
  Correlation betweenTumor mutation burden (TMB) and the efficacy
PK | Up to 2 years
  Pharmacokinetic profile in HCC patients of observed maximum plasma concentration
ADA | Up to 2 years
  Analysis of anti-drug antibody (ADA) during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer hospital, Beijing, China